CLINICAL TRIAL: NCT06722937
Title: The Collagen Factors of Rapid Progression of Keratoconus in Children: an Observational Cohort Study of the Physiological Parameter
Brief Title: The Collagen Factors of Rapid Progression of Keratoconus in Children.
Acronym: KCLD
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023KYPJ328
Record Dates: First submitted 2024-11-26; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Keratoconus
Keywords: keratoconus; pediatric; Corneal biomechanics; collagen
MeSH Terms: conditions — Keratoconus | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Venous blood DNA sequencing analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Keratoconus group of children
  Interventions: Other: Observation
- Keratoconus group of adult
  Interventions: Other: Observation
- Control group of children
  Interventions: Other: Observation
- Control group of adult
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observe the clinical natural changes of eye parameters of the subjects.

SUMMARY:
The purpose of this observational study was to understand the differences in clinical features and mechanisms of keratoconus between children and adults. The main questions it aimed to answer as follows: (1) to understand the characteristics of keratoconus in Chinese children. (2) to observe corneal stromal cells at the cytological level using in vivo corneal laser confocal microscopy and explore the pathogenesis.

DETAILED DESCRIPTION:
Keratoconus is a progressive and asymmetric corneal dilation disease, in which the cornea presents as a conical protrusion, leading to irregular astigmatism, progressive myopia, corneal thinning, and subsequent visual impairment. If left untreated, acute corneal edema may occur in the late stage, resulting in a sharp decline in vision. This disease is a binocular disease and can occur unilaterally first. The incidence rate of the general population is 1/2000. Most of the diseases described in the literature began in adolescence, and about 90% of the patients were diagnosed at the age of 10. Some literature reported that the youngest patient was 4 years old, and the disease generally remained stable until about 40 years old.

Currently, research on pediatric keratoconus mainly includes the prevalence and morphological characteristics, as well as the progression of corneal collagen cross-linking surgery. The younger onset age of KC is often associated with rapid progression and late stage disease diagnosis. Scholars have observed that 88% of children develop KC after one year of diagnosis, and advocate for early corneal collagen cross-linking treatment for these children's eyes. However, the reasons for the onset and progression of keratoconus in children at a young age are not yet clear.

Due to the young age of onset and unclear reasons for the progression of pediatric keratoconus in clinical practice, as well as insufficient research on pediatric keratoconus in recent years, the clinical characteristics of pediatric keratoconus are still lacking, and the pathogenesis of pediatric keratoconus is still unclear. Therefore, this study aims to compare pediatric keratoconus with adult keratoconus, extract the characteristics of pediatric keratoconus, and use a live corneal laser confocal microscope to observe the stromal cellular structure inside pediatric keratoconus, in order to provide some clinical reference for the pathological understanding of pediatric keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* ① Patients with keratoconus who visit the refractive clinic.

  1. The height of the posterior corneal surface is greater than 16 microns under the Pentacam corneal topography.
  2. ARTAve < 424 microns, ARTMax < 339 microns.
  3. Clinical non-inflammatory or traumatic corneal thinning and corneal astigmatism.

     * Aged between 10 and 50 years old, no gender restrictions.

       * Agree to accept and complete follow-up examinations on time. ④ I and my guardian understand and agree to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

* ① There is a history of contact lens wearing in the last four weeks.

  * poor fixation and can not cooperate with the examination. ③ History of eye trauma and surgery (including corneal collagen cross-linking surgery).

    * History of other related eye diseases: corneal disease, glaucoma, retinal choroid disease, etc..

      ⑤ severe eye diseases affecting imaging such as dry eye, conjunctivitis and pterygium.

      ⑥ Any systemic disease affecting eye morphology and refractive interstitium.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Consistently enrolled subjects aged between 10 and 50 years old with keratoconus and myopic astigmatism who visited the refractive clinic from April 2023 to April 2024
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-04-13 (Estimated); Study Completion 2025-04-13 (Estimated)

PRIMARY OUTCOMES:
Thinnest corneal thickness | 1 year
  Measurement of the thinnest point corneal thickness using the Three-Dimensional Anterior Segment Analyzer.
Kmax | 1 year
  Measurement of the maximum keratometry from the anterior corneal surface using the Pentacam Three-Dimensional Anterior Segment Analyzer.
ISV | 1 year
  Measurement of the index of surface variance of corneal front surface using the Pentacam Three-Dimensional Anterior Segment Analyzer.
IVA | 1 year
  Measurement of the index of vertical asymmetry of the corneal anterior surface using the Pentacam Three-Dimensional Anterior Segment Analyzer.
IHA | 1 year
  Measurement of the index of height asymmetry of the corneal anterior surface using the Pentacam Three-Dimensional Anterior Segment Analyzer.
IHD | 1 year
  Measurement of the index of height decentration the corneal anterior surface using the Pentacam Three-Dimensional Anterior Segment Analyzer.
CBI | 1 year
  Measurement of the corvis biomechanical index of cornea using the Corneal Biomechanical Analyzer.
TBI | 1 year
  Measurement of the tomographical biomechanical index of cornea using the Corneal Biomechanical Analyzer.
SPA1 | 1 year
  Measurement of the stiffness parameter at the first applanation of cornea using the Corneal Biomechanical Analyzer.
SSI | 1 year
  Measurement of the stress-strain index of cornea using the Corneal Biomechanical Analyzer.
Corneal stromal cell density | 1 year
  Measurement of the corneal stromal cell density using in vivo corneal confocal microscopy.
Mutations in collagen related genes | 1 year
  The expressions and mutations in collagen related genes(COL4A3, COL4A4 COL5A1, COL6A2, TGFBI, LOX, MMP9, TIMP1) using the DNA Sequencing Technology.

SECONDARY OUTCOMES:
Frame best corrected visual acuity | 1 year
  Measurement of best-corrected visual acuity of eye using visual charts.
Spherical power | 1 year
  Measurement of myopic refraction of eye using subjective refraction methods.
Cylindrical power | 1 year
  Measurement of astigmatism of eye using subjective refraction methods.
Axial length | 1 year
  Measurement of axial length of eye using IOL-Master 700.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center,Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
We will share our Study protocol, Statistical analysis plan, Informed consent form, Clinical study report.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting information will be permanently available (start date) on December 30, 2025.
Access Criteria: Any non-commercial scholars and institutions can apply to access the IPD and supporting information.

REFERENCES:
- See also: Registration information of this study in China — https://www.chictr.org.cn/